CLINICAL TRIAL: NCT04841304
Title: Cardiac Arrhythmia in Patients with End-Stage Renal Disease
Acronym: CADDY
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Herlev Hospital (Other); Steno Diabetes Center Copenhagen (Other); University of Copenhagen (Other); Hillerod Hospital, Denmark (Other); Holbaek Sygehus (Other)
Responsible Party: Principal Investigator, Bo Feldt-Rasmussen, Professor, Rigshospitalet, Denmark
Other Study IDs: H-20069767
Record Dates: First submitted 2021-03-26; First posted 2021-04-12 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: End Stage Renal Disease on Dialysis; Cardiac Arrhythmia; Diabetes Mellitus; Hypoglycemia
MeSH Terms: conditions — Arrhythmias, Cardiac; Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients receiving hemodialysis with diabetes: Patients receiving chronic hemodialysis with a diagnose of Type 1 diabetes or Type 2 diabetes (diagnosed according to the criteria of the World Health Organization) and receiving glucose-lowering treatment
  Interventions: Device: Loop recorder (Reveal LINQ, Medtronic); Device: Continuous Glucose Measurement (G6, Dexcom)
- Patients receiving hemodialysis without diabetes: Patients receiving chronic hemodialysis without diabetes (no known diagnosis of diabetes, and HbA1c < 48 mmol/mol at inclusion)
  Interventions: Device: Loop recorder (Reveal LINQ, Medtronic); Device: Continuous Glucose Measurement (G6, Dexcom)

INTERVENTIONS:
Device: Loop recorder (Reveal LINQ, Medtronic) — Implantation of a loop-recorder
Device: Continuous Glucose Measurement (G6, Dexcom) — Monitoring with a continuous glucose monitor

SUMMARY:
The study will examine the presence of cardiac arrhythmias in patients receiving hemodialysis and the role of diabetes, hypoglycemia and parameters related to uremia and the dialysis procedure.

The study is designed as a prospective cohort study with 18 months follow-up. 70 patients receiving chronic hemodialysis will be recruited and equipped with implantable loop recorders (ILR): 35 patients with diabetes and 35 patients without diabetes.

Data collection during the follow-up includes continuous monitoring of the heart rhythm by the ILR for the entire follow-up period, continuous glucose monitoring for 10 days every second month, and monthly collection of blood samples and dialytic parameters.

After the initial 18-month follow-up, heart rhythm monitoring will continue until the ILR battery runs out for those participants who wish to continue.

ELIGIBILITY:
Inclusion Criteria:

Patients with diabetes:

* Type 1 diabetes or Type 2 diabetes diagnosed according to the criteria of the World Health Organization
* Treated with glucose-lowering drugs at inclusion
* Receiving in-center maintenance hemodialysis for more than 3 months
* Age ≥ 18 years

Patients without diabetes:

* No known diagnosis of diabetes
* No previous treatment with glucose-lowering drugs
* HbA1c < 48 mmol/mol at screening
* Receiving in-center maintenance hemodialysis for more than 3 months
* Age ≥ 18 years

Exclusion Criteria:

For both groups:

* Cardiac pacemaker or implantable cardioverter defibrillator (ICD)
* Known permanent (chronic) atrial fibrillation
* History of sustained (> 30 seconds) ventricular tachycardia (more than 200 bpm) or ventricular fibrillation (note that ventricular premature beats is not considered an exclusion criterion)
* Known cardiac ion-channel disease (such as Long QT syndrome and Brugada syndrome)
* Not suitable for implantation (left-sided dialysis catheter or other condition expected to interfere with implantation)
* Previously complications in relation to wearing a CGM sensor, e.g. allergic reaction
* Inability to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 subjects receiving chronic hemodialysis therapy:
  * 35 subjects with diabetes
  * 35 subjects without diabetes
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Clinically significant arrhythmias | 18 months
  Presence of one of the items in the combined endpoint of clinically significant arrhythmias defined as:
  * Significant bradyarrhythmia (pause > 3 seconds or ≥ 4 beats at rate < 30 beats/min)
  * Ventricular tachycardia (lasting ≥ 16 beats at rate ≥ 150 beats/min)
  * Ventricular fibrillation

SECONDARY OUTCOMES:
Atrial fibrillation | 18 months
  Presence of atrial fibrillation (lasting ≥ 2 minutes)
Supraventricular tachycardia other than atrial fibrillation | 18 months
  Presence of supraventricular tachycardia other than atrial fibrillation (lasting ≥ 16 beats at rate ≥ 150 beats/min)
Time to clinically significant arrhythmias, atrial fibrillation, or supraventricular tachycardia, respectively | 18 months
  Time to clinically significant arrhythmias, atrial fibrillation, or supraventricular tachycardia, respectively
Characterization of arrhythmias in terms of onset | 18 months
  Characterization of arrhythmias in terms of onset
Characterization of arrhythmias in terms of duration | 18 months
  Characterization of arrhythmias in terms of duration
Characterization of arrhythmias in terms of ventricular rate | 18 months
  Characterization of arrhythmias in terms of ventricular rate
Episodes of hypoglycemia | 18 months
  Episodes of hypoglycemia <3.9 mmol/L (defined as sensor glucose below 3.9 mmol/L for ≥ 15 min)
Time in range | 18 months
  Time in range (percentage of time and amount of time with sensor glucose in range 3.9-10.0 mmol/L)
Time below range (<3.9 mmol/L) | 18 months
  Time below range (percentage time and amount of time with sensor glucose <3.9 mmol/L)
Time below range (<3.0 mmol/L) | 18 months
  Time below range (percentage of time and amount of time with sensor glucose <3.0 mmol/L)
Time above range (>10.0 mmol/L) | 18 months
  Time above range (percentage of time and amount of time with sensor glucose >10.0 mmol/L)
Time above range (>13.9 mmol/L) | 18 months
  Time above range (percentage of time and amount of time with sensor glucose >13.9 mmol/L)
Mean sensor glucose | 18 months
  Mean sensor glucose derived from continuous glucose monitoring
Glycemic variability | 18 months
  Glycemic variability (defined as coefficient of variation and standard deviation) derived from continuous glucose monitoring
Arrhythmia leading to the implantation of a cardiac implantable electronic device | 18 months
  Presence of any arrhythmia leading to the implantation of a cardiac implantable electronic device
Arrhythmia leading to a medical intervention | 18 months
  Presence of any arrhythmia leading to a medical intervention (defined as any change in prescribed medication)
Adverse events | 18 months
  Presence of adverse events, including procedure related adverse events
Sudden cardiac death | 18 months
  Sudden cardiac death
Cardiovascular death | 18 months
  Cardiovascular death
All-cause mortality | 18 months
  All-cause mortality

OTHER OUTCOMES:
Difference in arrhythmias between patients with diabetes and patients without diabetes | 18 months
  Difference in arrhythmias between patients with diabetes and patients without diabetes
Arrhythmias during hypoglycemia compared to euglycemia/hyperglycemia | 18 months
  Arrhythmias during hypoglycemia compared to euglycemia and hyperglycemia
The temporal distribution of arrhythmias in relation to hypoglycemic events | 18 months
  Arrhythmic events one hour prior to hypoglycemia, during hypoglycemia and one hour post hypoglycemia
Difference in glycemic characteristics between patients with and without diabetes | 18 months
  Difference in glycemic characteristics between patients with and without diabetes
Correlation between pre-dialysis blood samples and arrhythmias | 18 months
  Correlation between pre-dialysis blood samples and arrhythmias
Correlation between dialysis parameters and arrhythmias | 18 months
  Correlation between dialysis parameters (dialysate electrolyte concentrations and temperature) and arrhythmias
Correlation between a decline in systolic blood pressure during dialysis and arrythmias | 18 months
  Correlation between a decline in systolic blood pressure ≥20 mmHg during a dialysis session and arrythmias
Correlation between ultrafiltration rate and arrhythmias | 18 months
  Correlation between ultrafiltration rate and arrhythmias
The temporal distribution of arrhythmias in relation to dialysis sessions | 18 months
  Arrhythmic events eight hours prior to dialysis, during dialysis, eight hours post dialysis, and in the interval between dialysis sessions
Correlation between baseline clinical variables and arrhythmias | 18 months
  Correlation between baseline clinical variables (baseline demographic and comorbidity characteristics) and arrhythmias
Correlation between baseline residual diuresis and arrhythmias | 18 months
  Correlation between baseline residual diuresis and arrhythmias
Correlation between baseline electrocardiographic and echocardiographic markers and arrhythmias | 18 months
  Correlation between baseline electrocardiographic (assessed by 12-lead ECG) and echocardiographic markers (assessed by transthoracic echo) and arrhythmias
Correlation between heart rate variability, daytime and nighttime heart rate, physical activity, and risk of arrhythmias | 18 months
  Correlation between heart rate variability, daytime and nighttime heart rate, physical activity, and risk of arrhythmias

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Department of Nephrology, Rigshospitalet, Copenhagen
  - Department of Nephrology, Herlev Hospital, Herlev
  - Department of Nephrology, North Zealand Hospital, Hillerød
  - Department of Nephrology, Holbæk Sygehus, Holbæk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kofod DH, Diederichsen SZ, Bomholt T, Andersen MO, Andersen A, Mannheimer E, Rix M, Liem YS, Lindhard K, Hansen HP, Rydahl C, Lindhardt M, Brosen J, Schandorff K, Lange T, Norgaard K, Almdal TP, Svendsen JH, Feldt-Rasmussen B, Hornum M. Cardiac arrhythmia and hypoglycaemia among individuals with and without diabetes receiving haemodialysis (the CADDY study): a Danish multicentre cohort study. Diabetologia. 2025 Jun;68(6):1126-1139. doi: 10.1007/s00125-025-06388-5. Epub 2025 Feb 28. PMID 40019498
- [Derived] Kofod DH, Diederichsen SZ, Bomholt T, Orbaek Andersen M, Rix M, Liem Y, Lindhard K, Post Hansen H, Rydahl C, Lindhardt M, Schandorff K, Lange T, Norgaard K, Almdal TP, Svendsen JH, Feldt-Rasmussen B, Hornum M. Cardiac arrhythmia and hypoglycaemia in patients receiving haemodialysis with and without diabetes (the CADDY study): protocol for a Danish multicentre cohort study. BMJ Open. 2023 Oct 27;13(10):e077063. doi: 10.1136/bmjopen-2023-077063. PMID 37890966